CLINICAL TRIAL: NCT07186634
Title: Domain-Specific Appendix: OXYGEN
Brief Title: PeRiOperative Medicine Platform Trial
Acronym: PROMPT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Monash University (Other)
Collaborators: The Alfred (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-49324-130781
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Surgical Site Infection After Major Surgery; Anaesthesia; Major Complications; Quality of Recovery (QoR-15); Quality of Life
Keywords: Anaesthesiology, complications, oxygen, surgery; platform trial

STUDY DESIGN:
Intervention Model Description: conservative (≤30%), intermediate (50%), or liberal (80%) inspired oxygen concentration
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Liberal inspired oxygen (Active Comparator): FiO2 0.8; i.e. 80%
  Interventions: Drug: Liberal inspired oxygen
- Conservative inspired oxygen (Active Comparator): FiO2 ≤0.3 [30%]
  Interventions: Drug: Conservative inspired oxygen
- Intermediate inspired oxygen (Active Comparator): FiO2 0.5 [50%]
  Interventions: Drug: Intermediate inspired oxygen

INTERVENTIONS:
Drug: Liberal inspired oxygen — The concentration of Oxygen will differ according to the randomisation
  Arms: Liberal inspired oxygen
Drug: Conservative inspired oxygen — Conservative inspired oxygen
  Arms: Conservative inspired oxygen
Drug: Intermediate inspired oxygen — Intermediate inspired oxygen
  Arms: Intermediate inspired oxygen

SUMMARY:
Our specific aims are to investigate whether conservative (≤30%), intermediate (50%), or liberal (80%) inspired oxygen during and immediately after surgery: Aim 1: Reduces surgical site infections (SSIs or "wound infections") and other healthcare-associated infections (pneumonia and sepsis). Aim 2: Reduces a pooled composite of serious postoperative complications, leading to a faster and more complete recovery after surgery, and thus increases "days alive and at home up to 30 days after surgery" (DAH30). Primary hypothesis: Liberal (80%) oxygen concentration delivered with anesthesia in patients undergoing major surgery reduces the incidence of SSIs after surgery compared to conservative (≤30%) or intermediate (50%) oxygen concentration. Secondary hypothesis: Hyperoxia (50-80%) delivered with anesthesia in patients undergoing major surgery increases the incidence of pulmonary and other complications after surgery compared to conservative (≤30%) oxygen concentration, resulting in fewer Days At Home (DAH). PROMPT enrolls patients undergoing elective or semi-elective surgery.

DETAILED DESCRIPTION:
www.promptssi.org.au

ELIGIBILITY:
PROMPT - Inclusion Criteria:

* Adult patient (≥18 years of age at time of admission)
* Scheduled to undergo a surgical procedure involving a skin incision, with an expected duration of at least 2 hours, and a planned overnight hospital stay of at least 1 night (including, but not limited to, cardiac surgery, orthopedic surgery, obstetric, or gynecological surgery).

PROMPT - Exclusion Criteria:

* ASA physical status 5 (moribund, not expected to survive with or without an operation)
* Inability to provide informed consent
* Previous participation in PROMPT within the prior 30 days.

DSA 02 - PROMPT - Exclusion Criteria:

* ASA physical status 1 or 2
* Undergoing cardiac surgery
* Undergoing thoracic surgery if one-lung ventilation is required
* Currently suspected or proven infection
* Advanced lung disease requiring home oxygen therapy
* Previous bleomycin therapy
* Known or suspected pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7800 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection | 30 days
  A post operative infection that develops at the site of an operation, caused by bacteria entering the body through the surgical incision

SECONDARY OUTCOMES:
Health Care Associated Infections | 30 days
  pneumonia, blood stream infection and urinary tract infection
Quality of recovery | 3 and 30 days after surgery
  Quality of the individual's recovery post surgery - PROM. The scores of all 15 questions, with each item rated on a scale that results in a total score ranging from 0 (very poor recovery) to 150 (excellent recovery)
major postoperative complications | 30 days
  Description: A composite (and individually): Cardiovascular events (myocardial infarction, arterial or venous thrombosis, stroke, acute pulmonary edema, cardiogenic shock, new cardiac arrhythmia requiring treatment) Sepsis or septic shock (defined according to the Sepsis-3 definition)25 Respiratory complications - (i) pneumonia using US Centers for Disease Control criteria, (ii) Acute Respiratory Distress Syndrome using Berlin consensus definition, or (iii) the need for tracheal re-intubation and mechanical ventilation after extubation, and within 30 days after surgery OR mechanical ventilation for more than 24 h after surgery26 Unplanned intensive care unit (ICU) admission or readmission, defined as not anticipated preoperatively Acute kidney injury (based on the serum creatinine item of the Kidney Disease Improving Global Outcome criteria) Need for surgical re-intervention within 30 days after surgery Death within 30 days after surgery. Time Frame: 30 days
Mortality | 30 days
  All cause
EQ-5D-5L | 30 days
  Quality of life (EQ-5D-5L) at 30 days after index surgery. The resulting EQ-5D index score is a numerical value, with 1 representing full health, and scores less than 1 representing poorer health states, including negative values that indicate health states worse than death.
DAH 30 | 30 days
  Days alive and at home at 30 days (DAH30) after index surgery (reflecting the patient's primary aim of a healthy recovery, reduced hospital costs and the impact/severity of serious complications, and avoiding re-admission (often due to SSI).

OTHER OUTCOMES:
Cost Analysis | 30 days
  Direct health care costs at 30 days after index surgery Number of quality-adjusted life years (QALYs) at 30 days after index surgery Cost effectiveness measured as a cost per QALY.

CONTACTS AND LOCATIONS:
Overall Officials: Paul s Myles, DSc, Principal Investigator — Monash University; Trisha Peel, PhD, Principal Investigator — Monash University; Daniel Frei, PhD, Principal Investigator — Wellington Reginal Hospital
Locations (1):
- The Alfred, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
Dependent on Ethics Committee (IRB) approval, a clinically important hypothesis and valid protocol